CLINICAL TRIAL: NCT06350214
Title: Joint Association of Physical Activity and Dietary Quality With Survival Among US Cancer Survivors
Brief Title: Physical Activity and Nutrition in Cancer Survivors
Status: Completed | Type: Observational
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Lei Liu, Director, West China Hospital
Other Study IDs: #2005-06; #2011-17; #2018-01
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Cancer; Nutrition, Healthy; Physical Inactivity
MeSH Terms: conditions — Neoplasms; Sedentary Behavior | interventions — Exercise; Nutrition Assessment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: physical activity and nutrition assessment — Assessment of the physical activity and nutrition condition of cancer survivors.

SUMMARY:
This study aims to investigate the independent and combined associations between physical activity and nutrition condition with mortality among cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* Participants with history of cancers were included

Exclusion Criteria:

* Participants with missing cancer investigation, dietary recall, and incomplete follow-up information were excluded from this study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The data of this observational cohort study were extracted from six consecutive cycles of the Centers for Disease Control and Prevention's National Health and Nutrition Examination Survey (NHANES): including waves of 2007-2008, 2009-2010, 2011-2012, 2013-2014, 2015-2016, and 2017-2018. The NHANES database systematically gathered nationally representative health-related data on non-institutionalized general US civilians, utilizing a stratified, multistage probability sampling design.
Sampling Method: Probability Sample
Enrollment: 3100 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | Jan 1 2017 to Dec 31 2019
  To evaluate the overall survival of cancer survivors
Cause-specific mortality | Jan 1 2017 to Dec 31 2019
  To evaluate the cancer specific survival of cancer survivors

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Derived] Wei X, Min Y, Xiang Z, Zeng Y, Wang J, Liu L. Joint association of physical activity and dietary quality with survival among US cancer survivors: a population-based cohort study. Int J Surg. 2024 Sep 1;110(9):5585-5594. doi: 10.1097/JS9.0000000000001636. PMID 38874488